CLINICAL TRIAL: NCT06738498
Title: The Impact of Pre-Hospital and Hospital Delays on Myocardial Infarction Outcomes: A Prospective Study
Brief Title: Impact of Pre-Hospital and Hospital Delays on Myocardial Infarction Outcomes
Acronym: PHHD-MI
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241213A; 015 (Other: Nahrain Medical Research Collective (NMRC))
Record Dates: First submitted 2024-12-13; First posted 2024-12-17 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Myocardial Infarction (MI)
Keywords: Myocardial Infarction; Pre-Hospital Delay; Hospital Delay; Reperfusion Therapy; Patient Outcomes; Mortality; Time-to-Treatment; Cardiovascular Emergency
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this prospective observational study is to investigate the impact of pre-hospital and hospital delays on the outcomes of myocardial infarction (MI) patients admitted to Al-Kadhimiya Teaching Hospital, Baghdad.

The main questions it aims to answer are:

How do pre-hospital delays (e.g., patient transport and first medical contact) affect clinical outcomes such as mortality, complication rates, and recovery time in MI patients? What is the influence of hospital-related delays (e.g., time to intervention or reperfusion therapy) on the prognosis of MI patients?

Participants will:

Be monitored for the time elapsed from symptom onset to first medical contact and subsequent time intervals during hospital care.

Have their clinical outcomes, including in-hospital mortality, length of stay, and post-intervention complications, recorded and analyzed.

DETAILED DESCRIPTION:
Myocardial infarction (MI) continues to be one of the leading causes of cardiovascular mortality globally, with outcomes highly dependent on the timeliness of treatment. Early reperfusion therapy is crucial for reducing mortality and minimizing long-term complications such as heart failure and arrhythmias. The impact of delayed treatment, both in the pre-hospital and hospital phases, is well documented, with longer delays significantly worsening clinical outcomes, particularly in terms of mortality and myocardial damage. Meanwhile, recent studies indicate that time delays to care among patients with STEMI (ST-segment elevation myocardial infarction) exist universally, showing a worse situation in low- and middle-income countries than in high-income countries.

Hospital and pre-hospital delays are critical determinants of MI outcomes. Factors contributing to pre-hospital delays include patient-related issues, such as lack of recognition of symptoms, misinterpretation of their severity, and delays in decision-making, as well as external factors like geographical barriers to healthcare facilities and limited access to emergency medical services. Based on these findings, some national or regional programs have been initiated to reduce the delays by targeting at controlling these factors through educational campaigns, implementation of prehospital ECG, establishing regional collaborative networks, and these actions have turned out to be effective.

Additional contributing factors are also evident, including administrative inefficiencies, delays in diagnosis, and challenges in accessing specialized care such as percutaneous coronary intervention or thrombolysis. Evidence suggests that prolonged hospital delays increase the risk of adverse clinical outcomes, including higher rates of mortality and heart failure.

Previous studies have highlighted the significant influence of time on patient recovery. Research has shown that early reperfusion therapy, such as thrombolysis or percutaneous coronary intervention, can significantly improve patient survival and reduce the risk of long-term complications. However, despite extensive global studies, there is limited research that focuses on the unique delays encountered in Middle Eastern and low-resource settings like Iraq. The healthcare challenges in these regions, including access to timely emergency services and hospital readiness, require further investigation to provide actionable insights.

In Iraq, particularly in Baghdad, the impact of pre-hospital and hospital delays on MI outcomes remains underexplored. While cardiovascular diseases, including MI, are prevalent, the healthcare system faces significant challenges, such as limited public awareness, inadequate pre-hospital care, and hospital system constraints. These factors may contribute to substantial delays in MI treatment, but their specific impact on patient outcomes has not been well studied. This research aims to fill this gap by conducting a prospective observational study at Al-Kadhimiya Teaching Hospital in Baghdad, assessing the extent of pre-hospital and hospital delays in the management of MI and their correlation with clinical outcomes. The study seeks to identify critical delays and propose recommendations for improving the timeliness of MI care in Iraq.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provide informed consent (or a legal representative provides consent if the patient is unable to do so).
* Patients who undergo reperfusion therapy, such as thrombolysis or percutaneous coronary intervention (PCI).
* Patients admitted to Al-Kadhimiya Teaching Hospital within 12 hours of symptom onset.

Exclusion Criteria:

* Patients with non-acute myocardial infarction (e.g., stable angina, prior MI).
* Patients with severe comorbidities (e.g., advanced cancer, end-stage renal disease) that may complicate outcome assessments or interfere with treatment protocols.
* Patients who are transferred to another facility before reperfusion therapy is initiated.
* Pregnant women or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients aged 18 years and older who are diagnosed with acute myocardial infarction (MI), either STEMI or NSTEMI, confirmed by clinical symptoms, electrocardiogram (ECG), and elevated cardiac biomarkers (e.g., troponin). Participants will be admitted to Al-Kadhimiya Teaching Hospital within 12 hours of symptom onset and will undergo reperfusion therapy, such as thrombolysis or percutaneous coronary intervention (PCI).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
In-hospital Mortality | Up to discharge, an average of 7 days
  percentage of patients who die during hospitalization following myocardial infarction.

SECONDARY OUTCOMES:
Time-to-Reperfusion Therapy | Pre-Hospital Delay: Average of 4 hours from symptom onset to first medical contact. Hospital Delay: Average of 2 hours from hospital admission to the initiation of reperfusion therapy.
  The time (in minutes) from symptom onset to the initiation of reperfusion therapy (e.g., thrombolysis or percutaneous coronary intervention).
Length of Hospital Stay | Up to discharge, an average of 7 days
  The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge.
Major Adverse Cardiac Events (MACE) | Up to discharge, an average of 7 days
  Includes recurrent myocardial infarction, heart failure, and arrhythmias occurring during hospitalization.
Complication Rate | Up to discharge, an average of 7 days
  The proportion of patients developing complications related to delays in treatment (e.g., cardiogenic shock, ventricular rupture).

CONTACTS AND LOCATIONS:
Overall Officials: Aws Al-Rubaye Lecturer, Internal Medicine, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shehab A, AlHabib KF, Bhagavathula AS, Hersi A, Alfaleh H, Alshamiri MQ, Ullah A, Sulaiman K, Almahmeed W, Al Suwaidi J, Alsheikh-Ali AA, Amin H, Al Jarallah M, Salam AM. Clinical Presentation, Quality of Care, Risk Factors and Outcomes in Women with Acute ST-Elevation Myocardial Infarction (STEMI): An Observational Report from Six Middle Eastern Countries. Curr Vasc Pharmacol. 2019;17(4):388-395. doi: 10.2174/1570161116666180315104820. PMID 29542414
- [Background] Murray CJ, Lopez AD. Alternative projections of mortality and disability by cause 1990-2020: Global Burden of Disease Study. Lancet. 1997 May 24;349(9064):1498-504. doi: 10.1016/S0140-6736(96)07492-2. PMID 9167458
- [Background] GBD 2015 Mortality and Causes of Death Collaborators. Global, regional, and national life expectancy, all-cause mortality, and cause-specific mortality for 249 causes of death, 1980-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1459-1544. doi: 10.1016/S0140-6736(16)31012-1. PMID 27733281
- [Result] Ladwig KH, Fang X, Wolf K, Hoschar S, Albarqouni L, Ronel J, Meinertz T, Spieler D, Laugwitz KL, Schunkert H. Comparison of Delay Times Between Symptom Onset of an Acute ST-elevation Myocardial Infarction and Hospital Arrival in Men and Women <65 Years Versus >/=65 Years of Age.: Findings From the Multicenter Munich Examination of Delay in Patients Experiencing Acute Myocardial Infarction (MEDEA) Study. Am J Cardiol. 2017 Dec 15;120(12):2128-2134. doi: 10.1016/j.amjcard.2017.09.005. Epub 2017 Sep 18. PMID 29122276
- [Result] Peng YG, Feng JJ, Guo LF, Li N, Liu WH, Li GJ, Hao G, Zu XL. Factors associated with prehospital delay in patients with ST-segment elevation acute myocardial infarction in China. Am J Emerg Med. 2014 Apr;32(4):349-55. doi: 10.1016/j.ajem.2013.12.053. Epub 2014 Jan 3. PMID 24512889
- [Result] Naegeli B, Radovanovic D, Rickli H, Erne P, Seifert B, Duvoisin N, Pedrazzini G, Urban P, Bertel O. Impact of a nationwide public campaign on delays and outcome in Swiss patients with acute coronary syndrome. Eur J Cardiovasc Prev Rehabil. 2011 Apr;18(2):297-304. doi: 10.1177/1741826710389386. Epub 2011 Feb 11. PMID 21450676
- [Result] Park YH, Kang GH, Song BG, Chun WJ, Lee JH, Hwang SY, Oh JH, Park K, Kim YD. Factors related to prehospital time delay in acute ST-segment elevation myocardial infarction. J Korean Med Sci. 2012 Aug;27(8):864-9. doi: 10.3346/jkms.2012.27.8.864. Epub 2012 Jul 25. PMID 22876051
- [Result] Sullivan AL, Beshansky JR, Ruthazer R, Murman DH, Mader TJ, Selker HP. Factors associated with longer time to treatment for patients with suspected acute coronary syndromes: a cohort study. Circ Cardiovasc Qual Outcomes. 2014 Jan;7(1):86-94. doi: 10.1161/CIRCOUTCOMES.113.000396. Epub 2014 Jan 14. PMID 24425697
- [Result] Lee SH, Kim HK, Jeong MH, Lee JM, Gwon HC, Chae SC, Seong IW, Park JS, Chae JK, Hur SH, Cha KS, Kim HS, Seung KB, Rha SW, Ahn TH, Kim CJ, Hwang JY, Choi DJ, Yoon J, Joo SJ, Hwang KK, Kim DI, Oh SK; KAMIR Investigators. Pre-hospital delay and emergency medical services in acute myocardial infarction. Korean J Intern Med. 2020 Jan;35(1):119-132. doi: 10.3904/kjim.2019.123. Epub 2019 Nov 28. PMID 31766823
- [Result] George L, Ramamoorthy L, Satheesh S, Saya RP, Subrahmanyam DK. Prehospital delay and time to reperfusion therapy in ST elevation myocardial infarction. J Emerg Trauma Shock. 2017 Apr-Jun;10(2):64-69. doi: 10.4103/0974-2700.201580. PMID 28367010
- [Result] De Luca G, Suryapranata H, Ottervanger JP, Antman EM. Time delay to treatment and mortality in primary angioplasty for acute myocardial infarction: every minute of delay counts. Circulation. 2004 Mar 16;109(10):1223-5. doi: 10.1161/01.CIR.0000121424.76486.20. Epub 2004 Mar 8. PMID 15007008